CLINICAL TRIAL: NCT01440517
Title: An Open-Label, Multicenter, Proof of Concept, Phase 2 Study Evaluating the Results of Tc99m-Maraciclatide Scintigraphy in Subjects With Diabetes Mellitus (DM) and Heart Failure With Preserved Left Ventricular Ejection Fraction (HFPEF)
Brief Title: Results of Tc99m-Maraciclatide Scintigraphy in Subjects With Diabetes Mellitus and Heart Failure With Preserved Left Ventricular Ejection Fraction
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Subject Recruitment
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-078-101
Record Dates: First submitted 2011-09-22; First posted 2011-09-26 (Estimated); Results first posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-01

CONDITIONS: Diabetes Mellitus; Heart Failure
Keywords: CE-MRI - Contrast-enhanced magnetic resonance imaging; DM - Diabetes mellitus; EKG - Echocardiography; HFPEF - Heart failure preserved left ventricular ejection fraction; LVEF - Left Ventricular Ejection Fraction
MeSH Terms: conditions — Diabetes Mellitus; Heart Failure | interventions — NC100692; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tc99m-Maraciclatide (Experimental)
  Interventions: Drug: Tc99m-Maraciclatide

INTERVENTIONS:
Drug: Tc99m-Maraciclatide — Freeze-dried powder Kit for the preparation of Maraciclatide (99mTc) Injection
  Other Names: Maraciclatide (99mTc) Injection

SUMMARY:
The purpose of this study is to evaluate the results of 99mTc maraciclatide scintigraphy in diabetic subjects with HFPEF. A maximum of 20 subjects with Diabetes Mellitus (DM) and Heart Failure With Preserved Left Ventricular Ejection Fraction (HFPEF) will be enrolled and imaged with 99mTc maraciclatide. In addition, a maximum of 10 subjects with DM and diastolic dysfunction but no diagnosis of heart failure (HF) will be enrolled and imaged with 99mTc-maraciclatide.

ELIGIBILITY:
Inclusion Criteria:

* The subject is between 18 and 80 years of age.
* The subject was diagnosed with DM type 2 based upon accepted clinical criteria and currently takes at least one diabetes medication.
* For HF subjects: The subject was diagnosed with HF with preserved EF within the previous 1 year, at which time LVEF was determined to be ≥45%.
* For comparison subjects: The subject was determined to have diastolic dysfunction on EKG within the previous year and currently has no signs or symptoms of HF.
* The subject has been clinically stable for at least 7 days prior to the study imaging procedures (e.g., not experiencing continuing chest pain, hemodynamic instability, worsening HF symptoms, or clinically significant arrhythmia).

Exclusion Criteria:

* The subject had an acute myocardial infarction within the past 30 days.
* The subject had a cardiac revascularization (e.g., percutaneous transluminal coronary angiography [PTCA], percutaneous coronary intervention (PCI), or coronary artery bypass graft [CABG]) within the past 30 days.
* The subject has severe renal dysfunction.
* The subject is claustrophobic or has a movement disorder that prevents him/her from lying still in a supine position for up to 20 minutes at a time.
* The subject has participated in a research study using ionizing radiation in the previous 12 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Jacobson, MD, Study Director — GE Healthcare
Locations (1):
- GE Healthcare, Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Tc99m-Maraciclatide Injection: The nominal activity of a single administration of Tc88m maraciclatide was 925 megabecquerels (MBq) (25 millicures).
Period: Overall Study
Arm/Group | Tc99m-Maraciclatide Injection
Started | 5
Completed | 4
Not Completed | 1
Not completed — Subject withdrawn prior to dosing | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tc99m-Maraciclatide Injection
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Evidence of Active Myocardial Angiogenesis/Remodeling
Description: Due to the lack of subject enrollment, efficacy data were not analyzed.
Time Frame: Time zero equals the date of contrast imaging and for up to 24 hours for safety monitoring post contrast administration.
Population: Due to the lack of subject enrollment, efficacy data were not analyzed.
Arm/Group | Tc99m-Maraciclatide Injection
Number analyzed (Participants) | 0

2. Secondary Outcome: Uptake of 99mTc-maraciclatide Agent in Diabetic Subjects With Heart Failure With Preserved Left Ventricular Fraction and Subjects With Diabetes Mellitus and Asymptomatic Diastolic Dysfunction
Description: Due to the lack of subject enrollment, efficacy data were not analyzed.
Time Frame: Time zero equals the date of contrast imaging and for up to 24 hours for safety monitoring post contrast administration.
Population: Due to the lack of subject enrollment, efficacy data were not analyzed.
Arm/Group | Tc99m-Maraciclatide Injection
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Tc99m-Maraciclatide Injection
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 2/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tc99m-Maraciclatide Injection (N=4)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Diabetes Mellitus-Inadequate Control (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No